CLINICAL TRIAL: NCT06515080
Title: Physiological Monitoring in the OR; Predicting Outcomes Using Infra-red SEnsors, a Feasibility Study.
Brief Title: Predicting Outcomes Using Infra-red SEnsors, a Feasibility Study.
Acronym: PORPOISE-F
Status: Not yet recruiting | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: The University of Western Australia (Other); University of Sao Paulo (Other); Universitair Ziekenhuis Brussel (Other); Uppsala County Council, Sweden (Other Government); Istituto Giannina Gaslini (Other)
Responsible Party: Sponsor
Other Study IDs: PORPOISE Feasibility
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: General Anesthetic Drug Adverse Reaction
Keywords: regional oxygen saturation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children/Anesthesia
  Interventions: Diagnostic Test: Near Red Infrascopy

INTERVENTIONS:
Diagnostic Test: Near Red Infrascopy — Monitor of regional cerebral oxygen saturation

SUMMARY:
The aim of this study is to investigate if it is feasible to use a protocol in which avoiding oxygen desaturation in the brain during general anaesthesia can reduce the risk of negative postoperative behavior changes in children.

We will recruit children from at least five centres around the world for this feasibility study. Brain oxygenation will be monitored with Near Red Infrascopy (NIRS) which is like a saturation monitor placed on the forehead of the child during anesthesia. The anesthesia is done as per routine, but we will ask the anesthesiologist to record what actions they took when there were signs of decreasing oxygen saturation in the brain. We will also ask the parents to fill in a questionnaire with 27 questions about changes in their child's behavior 7 days after the operation.

DETAILED DESCRIPTION:
This project will investigate the potential effect of a protocol, targeted at counteracting cerebral desaturation during anaesthesia, with the aim of reducing negative post-operative changes in children. Negative post-operative changes (NPOBC) represent a surrogate outcome for neurocognitive damage associated with hemodynamic changes during general anaesthesia. This is a feasibility study that will examine anaesthesia team´s reactions to changes in (1) regional cerebral oxygen saturation (crSO2) (2) systemic hypotension or hypoxaemia, while also reporting any technical issues with data acquisition. We will also estimate the incidence of negative post-operative changes and explore any association with reduced crSO2 in our patient population compared with previous international data. Specifically, this feasibility study will provide data for the robust design and power analysis of a large-scale, randomised interventional trial in children undergoing anaesthesia, with the utilisation of a protocol targeting cerebral oxygen desaturation vs a control group of standard care with no access to crSO2 monitoring.

Methods At least 500 children of ages 6 months - 59 months will be recruited from at least 5 centers around the world. Besides routine monitoring, cerebral regional oxygen saturation (crsO2 will be monitored throughout the procedure.

Primary outcome The primary outcome is the feasibility of successful data collection of crO2, physiological and PHBQ data in a larger population over multiple international sites. This includes the incidence of technical problems with NIRS monitoring and the parental noncompliance with PHBQ reporting will be determined.

Secondary outcomes:

* The incidence of reduced crSO2 below baseline (more than 10%)
* The area under the curve (AUC) of reduced crSO2 below baseline
* The incidence of negative postoperative behaviour changes as determined by the PHBQ administered on day 7 & 30 following surgery.
* A set of threshold values for and form of interventions to restore cr02 and/or mean arterial blood pressure (Actions may include any of the following interventions fluid bolus, vasoactive agents, Trendelenburg position, adjustment of anaesthetic dose, and change of ventilation settings)
* The incidence of negative post-operative behavioural change and the extent of any association with the AUC of crSO2 below baseline

ELIGIBILITY:
Inclusion Criteria:

* Children scheduled for both elective and non-elective, non-cardiac surgical procedures under general anaesthesia.

Exclusion Criteria:

* age < 6 months or ≥ 59 months

  * procedures requiring < 30 minutes of general anaesthesia
  * imaging procedures
  * procedures involving neurosurgery, oncology or burns
  * procedures involving significant pain lasting for more than 1 week on average (e.g. tonsillectomies, major orthopaedic surgery)
  * other procedures that limit access to the forehead
  * children that are on supplemental oxygen, are sedated or intubated at the time of inclusion
  * children with severe developmental delay
  * procedures with planned postoperative intensive care or hospital stay > 3 days

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children undergoing routine general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
the incidence of technical problems with NIRS monitoring and the parental noncompliance with PHBQ reporting. Checklist | From the beginning of the anesthesia until 30 days postoperatively
  The primary outcome is the feasibility

SECONDARY OUTCOMES:
CrsO2 | From immediately before anesthesia induction until a few minutes after extubating up to 10 minutes
  Cerebral regional oxygen saturation monitored with NIRS
Negative postoperative behavior changes (NPOBC) | 7 to 30 days postoperatively
  Negative postoperative behavior changes detected by asking the parents to report changes of behavior assessed with the Post Hospitalization Behavior Questionnaire (PHBQ) at day 7 and day 30 postop

CONTACTS AND LOCATIONS:
Overall Officials: Peter Frykholm, M.D., Ph.D., Principal Investigator — Uppsala University
Locations (5):
- Perth Children´s Hospital, Perth, Western Australia, Australia
- Universitet Brussel, Brussels, Belgium
- University of Sao Paolo, São Paulo, Brazil
- Istituto Gaslini, Genova, Italy
- Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spaeder MC, Keller JM, Sawda CN, Surma VJ, Platter EN, White DN, Smith CJ, Harmon WG. Implementation of a Regional Oxygen Saturation Thought Algorithm and Association with Clinical Outcomes in Pediatric Patients Following Cardiac Surgery. Pediatr Cardiol. 2023 Apr;44(4):940-945. doi: 10.1007/s00246-022-03071-z. Epub 2022 Dec 13. PMID 36512036
- [Background] Gomez-Pesquera E, Poves-Alvarez R, Martinez-Rafael B, Liu P, Alvarez J, Lorenzo-Lopez M, Fierro I, Gomez-Sanchez E, Heredia-Rodriguez M, Gomez-Herreras JI, Tamayo E. Cerebral Oxygen Saturation and Negative Postoperative Behavioral Changes in Pediatric Surgery: A Prospective Observational Study. J Pediatr. 2019 May;208:207-213.e1. doi: 10.1016/j.jpeds.2018.12.047. Epub 2019 Feb 6. PMID 30737038
- [Background] McCann ME, de Graaff JC, Dorris L, Disma N, Withington D, Bell G, Grobler A, Stargatt R, Hunt RW, Sheppard SJ, Marmor J, Giribaldi G, Bellinger DC, Hartmann PL, Hardy P, Frawley G, Izzo F, von Ungern Sternberg BS, Lynn A, Wilton N, Mueller M, Polaner DM, Absalom AR, Szmuk P, Morton N, Berde C, Soriano S, Davidson AJ; GAS Consortium. Neurodevelopmental outcome at 5 years of age after general anaesthesia or awake-regional anaesthesia in infancy (GAS): an international, multicentre, randomised, controlled equivalence trial. Lancet. 2019 Feb 16;393(10172):664-677. doi: 10.1016/S0140-6736(18)32485-1. Epub 2019 Feb 14. PMID 30782342
- [Background] Jevtovic-Todorovic V, Useinovic N. Early exposure to general anaesthesia and increasing trends in developmental behavioural impairments: is there a link? Br J Anaesth. 2023 Aug;131(2):208-211. doi: 10.1016/j.bja.2023.04.005. Epub 2023 May 10. PMID 37173202